CLINICAL TRIAL: NCT01505348
Title: Effect of Fasting Versus Feeding on the Bone Metabolic Response to Running
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: QinetiQ Ltd (Industry)
Collaborators: Ministry of Defence, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: QQ-SP751
Record Dates: First submitted 2012-01-04; First posted 2012-01-06 (Estimated); Last update posted 2012-01-06 (Estimated); Status verified 2012-01

CONDITIONS: Feeding Patterns; Bone Resorption
Keywords: feeding patterns; aerobic exercise; osteoclasts
MeSH Terms: conditions — Feeding Behavior; Bone Resorption | interventions — Angptl4 protein, mouse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fasting (Experimental): Overnight fast
  Interventions: Other: Overnight fast
- Feeding (No Intervention): Normal breakfast

INTERVENTIONS:
Other: Overnight fast — Overnight fast from 21:00 h
  Other Names: Fasting
  Arms: Fasting

SUMMARY:
This study examined changes in bone metabolism (markers of bone turnover, calcium metabolism) with a bout of acute treadmill running preceded by either a single, mixed meal or an overnight fast.

DETAILED DESCRIPTION:
Ten physically active males aged 28 ± 4 y (mean ± 1SD) completed two, counterbalanced, 8 d trials. After 3 d on a standardised diet, participants performed 60 min of treadmill running at 65% VO2max on Day 4 following an overnight fast (FAST) or a standardised breakfast (FED). Blood samples were collected at baseline, before exercise, during exercise, for 3h after exercise and on four consecutive follow-up days (FU1-FU4). Plasma/serum were analysed for β CTX, P1NP, OC, bone ALP, PTH, ACa, PO4, OPG, cortisol, leptin and ghrelin.

ELIGIBILITY:
Inclusion Criteria:

* history of weight bearing exercise
* fasting vitamin D concentration of >30 nmol•L-1 and/or a fasting parathyroid hormone (PTH) concentration of <6.9 pmol•L-1.

Exclusion Criteria:

* smokers
* suffered a bone fracture in the previous 12 months
* musculoskeletal injury
* condition/medication known to affect bone metabolism

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2007-07; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Change in C-terminal telopeptide region of collagen type 1 (B-CTX) concentration from baseline | At 08:00 h (Baseline), 09:00 h, 09:30 h, and 10:15 h (Pre-exercise), after 30 and 60 min of exercise, after 1, 2, and 3 h of recovery and at 1, 2, 3 and 4 day post-exercise
  B-CTX is a specific marker of bone resorption. It's circulating concentration is altered by both exercise and feeding

SECONDARY OUTCOMES:
Change in parathyroid hormone (PTH) concentration from baseline | At 08:00 h (Baseline), 09:00 h, 09:30 h, and 10:15 h (Pre-exercise), after 30 and 60 min of exercise, after 1, 2, and 3 h of recovery and at 1, 2, 3 and 4 day post-exercise
  PTH is reported to induce both bone resorption and bone formation. It's circulating concentration is altered by both exercise and feeding.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan PR Scott, Ph.D, Principal Investigator — QinetiQ Ltd
Locations (1):
- QinetiQ Ltd, Farnborough, Hampshire, United Kingdom